CLINICAL TRIAL: NCT02725398
Title: Effect of Buscopan on Gastrointestinal Imaging Quality With Probe-based Confocal Laser Endomicroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Shuhui Liang, Associated Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: pCLE-BSP
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Gastrointestinal Imaging With pCLE
Keywords: Buscopan; probe-based confocal laser endomicroscopy; Imaging Quality
MeSH Terms: interventions — Butylscopolammonium Bromide; Scopolamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Buscopan group (Experimental): First to use standard white light to observe, to record spasm score, to observe the lesion.Buscopan (BSP, 20mg) is administered by endoscopic nurse, recorded blindly.
  Interventions: Drug: Buscopan
- Scopolamine group (Active Comparator): First to use standard white light to observe, to record spasm score, to observe the lesion.Scopolamine is administered by endoscopic nurse, recorded blindly.
  Interventions: Drug: Scopolamine
- physiological saline group (Placebo Comparator): First to use standard white light to observe, to record spasm score, to observe the lesion. Physiological saline is administered by endoscopic nurse, recorded blindly.
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Buscopan — Buscopan is administered by endoscopic nurse in the Buscopan group,and then recording the outcome measures.
  Other Names: Butylscopolammonium Bromide
  Arms: Buscopan group
Drug: Scopolamine — Scopolamine is administered by endoscopic nurse in the Scopolamine group,and then recording the outcome measures.
  Other Names: 654-2, in China
  Arms: Scopolamine group
Drug: physiological saline — Physiological saline is administered by endoscopic nurse in the physiological saline group,and then recording the outcome measures.
  Other Names: Sodium Chloride Physiological Solution; NS, normal saline
  Arms: physiological saline group

SUMMARY:
Gastrointestinal cancer has developed into a serious health problem in China. 80%-90% patients were detected at middle and later stage. The five-year survival rate for advanced cancer patients is less than 10%. The main reason of the bad clinical diagnosis and treatment is that the present technical method is difficult to achieve early diagnosis. Endoscopy with biopsy is still the main method for confirming gastrointestinal cancer. But it is limited to identify early tumors and it leads to the low diagnostic rate of early tumors and the poor overall therapeutic effect.

Confocal laser endoscopy (CLE) can obtain pathologic information of lesion in real time and improve the diagnostic rate of early tumors. Probe-based confocal laser endomicroscopy(pCLE) is a new technology recently. Since its laser probe is applicable to all conventional endoscopes, pCLE greatly increased its clinical application. However, gastrointestinal motility has greatly influence on pCLE imaging quality and inspection effect owing to the poor stability of the small probe manipulation. Scopolamine (654-2, in China) is clinically used to inhibit bowel peristalsis, but its effect is still not ideal and its side effects are common.

DETAILED DESCRIPTION:
Buscopan can more effectively relieve gastrointestinal spasm, and its side effects is fewer. It has been reported that Buscopan can more effectively relieve gastrointestinal spasm, facilitate scope insertion and improve patients' comfort during endoscopy.Buscopan may make the endoscopic physicians to observe easily and effectively improve the diagnostic rate. Buscopan may effectively inhibit duodenum motility and facilitate the ERCP operation.It has not been reported in the literature whether Buscopan can be used on pCLE examination to improve imaging quality and the detection accuracy of the lesion.

Hence, the investigators plan to develop a prospective, double-blind, randomized, controlled study, the effect of Buscopan on gastrointestinal imaging quality and diagnosis accuracy with probe-based confocal laser endomicroscopy, in order to confirm the practical application value of Buscopan in pCLE examination.

Patient selection, grouping, and operating process:

Subjects were selected based on the inclusion and exclusion criterion from the volunteers eligible for this trial who are inpatient or outpatient applying for pCLE examination in the endoscopy center of Xijing Digestive Disease Hospital. Patients were divided into three groups: Buscopan (BSP), Scopolamine (654-2) and physiological saline (NS) control group, according to the ratio of 1:1:1. Operators were blind to random grouping,and patients were unclear to accept Buscopan, 654-2 or NS drugs before operation. All endoscopy operation should be completed by clinical experienced endoscopists (WKC or LSH) by using gastroscopy、 colonoscopy and enteroscopy, respectively GIF-H260、CF-H260、SIF-260 (Olympus Medical Systems, Tokyo, Japan).

Operating process: Preoperative preparation are basically the same to conventional endoscopy.Patients ingested mucosal surface anesthesia and defoaming agent 30 minutes before endoscopy,and accepted the fluorescein sodium allergy test intravenously (2%, 1 ml) 20 minutes before endoscopy, established venous pathway. Negative patients could accept pCLE examination. First to use standard white light to observe, to record spasm score,to observe the lesion. It is administered by endoscopic nurse which is respectively Buscopan (BSP, 20mg), Scopolamine (654-2,10mg), physiological saline (NS), recorded blindly. Then to inject 10% fluorescein sodium 5ml (Guangzhou Baiyun Shan Ming Xing Pharmaceutical Co., Ltd.) intravenously,to start button to scan by pCLE. To scan in the order of the back of endoscopy,to indicate each observation position by pCLE, to do targeted biopsy by pCLE if met lesion. During the examination,spasm scores (2 minutes,20 minutes after administering drug) and operation time were recorded. Visual analogue scale (visual field stability and patient comfort) level was given after the examination. To record whether related complications happen and positively process. To evaluate the quality of each imaging according to Kiesslich pCLE image quality analysis method and diagnostic accuracy combining with the pathologic diagnosis(through the target biopsy, pathological examination, comparative calculation).

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 years
* Sex unlimited
* Patients who were suspected or previous gastrointestinal disease
* Screening outpatients
* Other patients who are willing to accept the case of CLE

Exclusion Criteria:

* Patients with severe heart or pulmonary disease which is not suitable for endoscopic examination
* Pregnant or lactating female
* Patients who were allergic to contrast medium or clinical drug
* Higher blood risk of esophageal varices
* Patients who were known or suspected gastrointestinal stenosis or obstruction
* Patients who had prostatic hypertrophy, or glaucoma and so on
* Without patient's consent
* Others who can not cooperate with endoscopic examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
high quality image ratio | up to 3 years

SECONDARY OUTCOMES:
spasm score | 3 years
  the rate which spasm score decline was significant (spasm score decline two points before and after the drug)
diagnosis accuracy rate | 3 years
  the rate of participants among which the pCLE diagnosis agree with the pathologic diagnosis
scale value of patient' comfort degree assessed by using visual analogue scale (VAS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, M.D., Prof., Study Director — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes